CLINICAL TRIAL: NCT07216365
Title: Caffeine Optimization for Oxygen Saturation Index in ELBW Infants (COFIE Trial)
Brief Title: Caffeine Optimization for Oxygen Saturation Index in ELBW Infants
Acronym: COFIE trail
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Stephanie Vachon, Assistant Professor - Department of Pediatrics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00000000
Record Dates: First submitted 2025-09-05; First posted 2025-10-14 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-10

CONDITIONS: Neonatal Apnea; Infants
MeSH Terms: interventions — caffeine citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Dose Caffeine Arm (Experimental): Infants randomized to the high dose caffeine arm will receive an initial standard loading dose of 20 mg/kg caffeine citrate. Beginning at 7 days of life, they will receive a maintenance dose of 10 mg/kg/day caffeine citrate. Dose escalation may be performed at the discretion of the clinical team, with a maximum maintenance dose of 12.5 mg/kg/day if clinically indicated. Caffeine will be administered IV or PO at a 1:1 ratio and prepared in a blinded fashion.
  Interventions: Drug: Caffeine Citrate
- Standard Dose Caffeine Arm (Active Comparator): Infants randomized to the standard dose caffeine arm will receive an initial loading dose of 20 mg/kg caffeine citrate. Beginning at 7 days of life, they will receive a maintenance dose of 5 mg/kg/day. Dose escalation may occur at the discretion of the clinical team, with a maximum maintenance dose of 7.5 mg/kg/day. Caffeine will be administered IV or PO at a 1:1 ratio and prepared in a blinded fashion.
  Interventions: Drug: Caffeine Citrate

INTERVENTIONS:
Drug: Caffeine Citrate — High Dose Group:
  Caffeine citrate administered as a 20 mg/kg loading dose followed by a 10 mg/kg/day maintenance dose starting at 7 days of life. Dose escalation up to 12.5 mg/kg/day may be performed based on clinical indications. The drug is administered either intravenously or orally in a blinded fashion.
  Standard Dose Group:
  Caffeine citrate administered as a 20 mg/kg loading dose followed by a 5 mg/kg/day maintenance dose starting at 7 days of life. Dose escalation up to 7.5 mg/kg/day may be performed based on clinical indications. The drug is administered either intravenously or orally in a blinded fashion.

SUMMARY:
The goal of this clinical trial is to determine whether a higher dose of caffeine citrate can improve breathing and reduce health complications in extremely premature infants, specifically those born before 28 weeks of pregnancy, known as ELGAN infants. These babies often struggle with breathing due to underdeveloped lungs, and caffeine is commonly used to help support their respiratory function. However, the most effective and safest dose has not yet been clearly established.

The study aims to answer two main questions: Does a higher maintenance dose of caffeine (10 mg/kg) lead to better oxygenation, as measured by the Oxygen Saturation Index (OSI), compared to the standard dose (5 mg/kg)? And does the higher dose reduce the risk of serious complications such as lung disease, brain injury, or death-without causing more side effects like fast heart rate, high blood pressure, or poor growth?

To answer these questions, researchers will compare two groups of infants: one receiving the high-dose caffeine treatment and the other receiving the standard dose. This comparison will help determine if the higher dose leads to better outcomes without increased risk.

Participants will begin caffeine treatment once they have regained their birth weight and are at least seven days old. They will be randomly assigned to receive either the high or standard caffeine dose and will be followed until caffeine is stopped or they are discharged from the hospital. During this time, researchers will monitor each infant's oxygenation levels, need for breathing support, signs of common complications, growth and feeding progress, and any side effects. Before discharge, each infant's motor development will also be assessed using a tool called the Test of Infant Motor Performance (TIMP).

This study could help define the most effective caffeine dosing strategy for supporting extremely premature infants and improving their short-term health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* URMC Inborn Newborn infants born with gestational age of 22 weeks 0 days - 27 weeks 6 days or infants OR ≥ 28 weeks with a birthweight < 1000 grams

Exclusion Criteria:

* Hepatic failure, spontaneous intestinal perforation, necrotizing enterocolitis, Anticipated major congenital or genetic anomalies, infants not anticipated to survive beyond 72 hours, infants with mothers that are non-English speaking or <18 years old at time of enrollment.

Ages: 0 Days to 27 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Average Oxygen Saturation Index (OSI) per Patient Over First 56 Days | From Randomization to Day 56 or Caffeine Discontinuation
  The OSI is calculated as (FiO₂ × MAP × 100) / SpO₂. The average OSI per patient will be calculated from randomization through the first 56 days or until caffeine is discontinued or the patient is discharged. Higher OSI values indicate worse oxygenation.
Total Duration of Respiratory Support | From Randomization to 1 year
  Total number of days each patient receives any respiratory support, including invasive ventilation, CPAP, or supplemental oxygen.
Total Incidence of Severe Bronchopulmonary Dysplasia (BPD) | From Randomization to 1 year
  Number of infants diagnosed with severe BPD based on NICHD criteria.
Total Incidence of Severe Intraventricular Hemorrhage or Periventricular Leukomalacia (IVH/PVL) | From Randomization to 1 year
  Number of infants diagnosed with severe IVH (Grade III/IV) or PVL based on cranial imaging.
Total Length of NICU Stay | Birth to 1 year
  Total number of days each infant remains in the NICU from birth until discharge.
Total Number of Infant Deaths | From Randomization to 1 year
  Number of infants who die before NICU discharge.
Total Test of Infant Motor Performance (TIMP) Score Prior to Discharge | Prior to NICU Discharge
  TIMP is a 42-item motor development assessment. Each item scores from 0 to 6. Total scores range from 0 to 252. Higher scores indicate better motor performance.
Total Duration of SpO₂ Below Threshold (Intermittent Hypoxia) | From Randomization through Day 56
  Cumulative minutes with SpO₂ below target threshold, derived from Neo-DReAMS repository.
Total Time with Heart Rate >180 bpm (Tachycardia) | From Randomization to 1 year
  Total minutes with heart rate exceeding 180 bpm recorded via monitor.
Total Growth Parameter Z-Scores (Length, Weight, Head Circumference) | From Randomization to 1 year
  Growth will be assessed using Fenton z-scores. Higher scores reflect better growth relative to gestational norms.
Total Osteopenia Markers (Alkaline Phosphatase, Calcium, Phosphorus) | From Randomization to 1 year
  Osteopenia assessed by abnormal lab values: alkaline phosphatase >500 IU/L, abnormal calcium or phosphorus. Abnormal values per infant will be summed.
Total Incidence of Hypertension (>95th Percentile) | From Randomization to 1 year
  Number of days with blood pressure >95th percentile for gestational age.
Total Time to Full Enteral Feeds | From Randomization to 1 year
  Days from birth until the infant reaches 120 mL/kg/day enteral nutrition.
Total Number of NPO Periods >24 Hours | From Randomization through NICU Discharge
  Number of times infant is NPO (nothing by mouth) for more than 24 hours.
Total Incidence of Necrotizing Enterocolitis (NEC) | From Randomization to 1 year
  Number of infants diagnosed with NEC (Bell's stage II or higher).
Total Incidence of Spontaneous Intestinal Perforation (SIP) | From Randomization to 1 year
  Number of infants with radiographically or surgically confirmed SIP.

IPD SHARING:
Plan to Share IPD: No